CLINICAL TRIAL: NCT07157956
Title: Phase I/II Clinical Study of CVL006 Combination Therapy in Advanced Solid Tumors
Brief Title: CVL006 Combination Therapy in Advanced Solid Tumors
Acronym: CVL006-T1002
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Convalife (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVL006-T1002
Record Dates: First submitted 2025-08-22; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; DLT; RP2D
MeSH Terms: interventions — Pemetrexed; Carboplatin; trastuzumab deruxtecan; enfortumab vedotin

STUDY DESIGN:
Intervention Model Description: This study is a multi-center, open-label, dose-escalation and dose-optimized phase I/II clinical trial. Objective: To determine the safety, tolerability, PK characteristics and preliminary efficacy data of CVL006 combined with pemetrexed + carboplatin/SKB264/ DS-8201a/ Enfortumab Vedotin in patients with advanced solid tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Arm 1.1 (Experimental): Patients with advanced solid tumors were enrolled in Arm1.1. The medication used was CVL006 combined with pemetrexed and carboplatin. Two dose groups were preset. The starting dose of CVL006 for DL1 was 10mg/kg (administered at Q2W or Q3W), and for DL2 (one dose higher than DL1). Pemetrexed + carboplatin was a fixed dose. Each dose group enrolled 3 to 6 patients, and Arm1.1 enrolled a total of 6 to 12 patients.
  Interventions: Drug: CVL006 combined with pemetrexed and carboplatin
- Arm 1.2 (Experimental): Patients with advanced solid tumors were enrolled in Arm1.2, and the medication used was CVL006 combined with SKB264. Two dose groups were preset. The starting dose of CVL006 for DL1 was 10mg/kg (administered at Q2W or Q3W), and for DL2 (one dose group higher than DL1). SKB264 was a fixed dose. Each dose group enrolled 3 to 6 patients, and Arm1.2 enrolled a total of 6 to 12 patients.
  Interventions: Drug: CVL006 in combination with SKB264
- Arm 1.3 (Experimental): Patients with advanced solid tumors were enrolled in Arm1.3, and the medication used was CVL006 combined with DS-8201a. Two dose groups were preset. The starting dose of CVL006 for DL1 was 10mg/kg (administered at Q2W or Q3W), and the dose for DL2 (one dose group higher than DL1). DS-8201a was a fixed dose. Each dose group enrolled 3 to 6 patients respectively, and Arm1.3 enrolled a total of 6 to 12 patients.
  Interventions: Drug: CVL006 in combination with DS-8201
- Arm1.4 (Experimental): Patients with advanced solid tumors were enrolled in Arm1.4 and treated with CVL006 combined with Enfortumab Vedotin. Two dose groups were preset. The starting dose of CVL006 for DL1 was 10mg/kg (administered at Q2W or Q3W), and the dose of DL2 (one dose group higher than DL1). Enfortumab Vedotin was a fixed dose. 3 to 6 patients were enrolled in each dose group, and 6 to 12 patients were enrolled in Arm1.4.
  Interventions: Drug: CVL006 in combination with Enfortumab Vedotin
- Arm2.1 (Experimental): NSCLC patients were enrolled in Arm2.1. The medication used was CVL006 combined with pemetrexed and carboplatin. 8 to 30 patients were enrolled.
  Interventions: Drug: CVL006 combined with pemetrexed and carboplatin
- Arm2.2 (Experimental): Patients with EGFRm nsqNSCLC were enrolled in Arm2.2. The medication used was CVL006 combined with pemetrexed and carboplatin. 8 to 30 patients were enrolled.
  Interventions: Drug: CVL006 combined with pemetrexed and carboplatin
- Arm2.3 (Experimental): Patients with malignant pleural mesothelioma were enrolled in Arm2.3. The medication used was CVL006 combined with pemetrexed and carboplatin. 8 to 30 patients were enrolled.
  Interventions: Drug: CVL006 combined with pemetrexed and carboplatin
- Arm2.4 (Experimental): Breast cancer patients were enrolled in Arm2.4, and the medication used was CVL006 combined with SKB264. 8 to 30 patients were enrolled.
  Interventions: Drug: CVL006 in combination with SKB264
- Arm2.5 (Experimental): Patients with EGFRm nsqNSCLC were enrolled under Arm2.5, with the medication being CVL006 combined with SKB264. 8 to 30 patients were enrolled.
  Interventions: Drug: CVL006 in combination with SKB264
- Arm2.6 (Experimental): Breast cancer patients were enrolled in Arm2.6, and the medication used was CVL006 combined with DS-8201a. 8 to 30 patients were enrolled.
  Interventions: Drug: CVL006 in combination with DS-8201
- Arm2.7 (Experimental): NSCLC patients were enrolled in Arm2.7. The medication used was CVL006 combined with DS-8201a. 8 to 30 patients were enrolled.
  Interventions: Drug: CVL006 in combination with DS-8201
- Arm2.8 (Experimental): Patients with adenocarcinoma of the stomach or gastroesophageal junction were enrolled under Arm2.8. The medication used was CVL006 combined with DS-8201a. 8 to 30 patients were enrolled.
  Interventions: Drug: CVL006 in combination with DS-8201
- Arm2.9 (Experimental): Patients with urothelial carcinoma were enrolled under Arm2.9. The medication used was CVL006 combined with Enfortumab Vedotin. 8t to 30 patients were enrolled.
  Interventions: Drug: CVL006 in combination with Enfortumab Vedotin

INTERVENTIONS:
Drug: CVL006 combined with pemetrexed and carboplatin — CVL006 combined with pemetrexed and carboplatin
  Other Names: CVL006（B006 Injection）、pemetrexed（Pemetrexed Disodium for Injection）、carboplatin（Carboplatin Injection）
  Arms: Arm 1.1; Arm2.1; Arm2.2; Arm2.3
Drug: CVL006 in combination with SKB264 — CVL006 in combination with SKB264
  Other Names: CVL006（B006 Injection）、SKB264（Sacituzumab tirumotecan）
  Arms: Arm 1.2; Arm2.4; Arm2.5
Drug: CVL006 in combination with DS-8201 — CVL006 in combination with DS-8201
  Other Names: CVL006（B006 Injection）、DS-8201a（Trastuzumab deruxtecan）
  Arms: Arm 1.3; Arm2.6; Arm2.7; Arm2.8
Drug: CVL006 in combination with Enfortumab Vedotin — CVL006 in combination with Enfortumab Vedotin
  Other Names: CVL006（B006 Injection）、Enfortumab Vedotin（Padcev）
  Arms: Arm1.4; Arm2.9

SUMMARY:
This study is a multi-center, open-label, dose-escalation and dose-optimized phase I/II clinical trial. Objective: To determine the safety, tolerability, PK characteristics and preliminary efficacy data of CVL006 combined with pemetrexed + carboplatin/SKB264/ DS-8201a/ Enfortumab Vedotin in patients with advanced solid tumors.

DETAILED DESCRIPTION:
1. Phase I Arm1.1 - Arm1.4: Dose escalation of CVL006 combined with pemetrexed + carboplatin/SKB264/ DS-8201a/ Enfortumab Vedotin: Dose escalation studies of CVL006 combined with pemetrexed + carboplatin/SKB264/DS-8201a/ Enfortumab Vedotin can be conducted simultaneously, with two dose groups preset for each combination: The starting Dose (Dose Level1 [DL1]) of CVL006 is 3mg/kg or more (the investigator and the sponsor can discuss and decide on a dose of 3mg or more based on more data from the Phase I monotherapy study), Q2W or Q3W administration, and DL2 (one dose group higher than DL1) dose. Arm1.1 to Arm1.4 Each cohort is expected to increase to 6 to 12 subjects. Based on the data such as safety, tolerability, efficacy and PK characteristics observed during the dose escalation process of each cohort, the researcher and the sponsor jointly decided whether to adopt the Backfill design, that is, to enroll additional patients in the confirmed safe low-dose group during the dose escalation process. And decide whether to explore other administration doses or frequencies (such as Q3W).
2. Phase II Dose optimization study In order to further evaluate the PK characteristics, safety and preliminary anti-tumor activity of CVL006 combined with pemetrexed + carboplatin/SKB264/ DS-8201a/ Enfortumab Vedotin, while the dose escalation trial of phase I was being conducted, Several dose groups that have passed the safety assessment during the DLT observation period will be selected to conduct the Phase II dose expansion study simultaneously. If, based on the obtained safety, tolerability, PK and efficacy information, the investigator and the sponsor discuss and decide on the choice of dose expansion and the specific number of cases to be increased. And whether a new dose needs to be added for dose expansion. Similarly, for each cohort with a new dose or a new administration frequency, the number of subjects in each group should be increased to 8-30 (subjects who previously used the same dose can be included).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old (including both ends), gender not limited;
2. Stage I Arm1.1, Arm1.2, Arm1.3 and Arm1.4: Locally advanced, recurrent or metastatic solid tumors confirmed by histology or cytology, with previous treatment failure.
3. Phase II Arm2.1, Arm2.2, Arm2.5 and Arm2.7: For NSCLC Arm2.1: Non-squamous, wild-type NSCLC Arm2.2: EGFRm nsqNSCLC Arm2.3: Malignant pleural mesothelioma Arm2.4: triple-negative breast cancer Arm2.5: EGFRm nsqNSCLC Arm2.6: breast cancer Arm2.7: NSCLC Arm2.8: adenocarcinoma of the stomach or gastroesophageal junction Arm2.9: urothelial carcinoma
4. All subjects must provide tumor tissue samples for PD-L1 testing: Tumor tissue samples should preferably be newly obtained tumor tissues. For subjects who cannot provide newly obtained tissues, tumor tissue samples archived within 3 years prior to the first study treatment can be provided. The sample type should be neutral formalin-fixed and paraffin-embedded [FFPE] tissue wax blocks or at least 6 unstained tumor tissue sections. If the number is less than 6 pieces, it is necessary to negotiate with the sponsor and only allow enrollment after obtaining consent.
5. ECOG overall performance status (PS) 0-1 point;
6. Predicted survival period ≥ 3 months;
7. According to the efficacy evaluation criteria for solid tumors (RECISTv 1.1), there is at least one measurable lesion;
8. Have sufficient bone marrow and organ function (no blood components and/or cell growth factors have been used within 14 days prior to the start of the study treatment) :

   Hemoglobin (HB) ≥ 90 g/L;

   • Neutrophil count (ANC) ≥1.5×109/L;

   Platelet count (PLT) ≥ 90×109/L;

   • Total bilirubin < 1.5×ULN (for subjects diagnosed with Gilbert syndrome, total bilirubin ≤ 3×ULN);
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN (for patients with liver metastasis, ALT and/or AST≤ 5×ULN);
   * Serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 60 mL/min (calculated according to the Cockcroft-Gault formula);
   * International normalized ratio (INR) and activated partial thromboplastin (APTT) time ≤1.5×ULN;
   * Qualitative urine protein ≤1+; Or the qualitative urine protein is ≥2+, and the 24-hour urine protein should be less than 1g
9. Fertile women must agree to abstain from sexual activity (avoiding heterosexual intercourse) or use effective contraceptive methods for at least six months from the date of signing the informed consent form until the last administration of the study drug. Moreover, the blood HCG test must be negative within 7 days before the start of the study treatment, and the patient must not be in the lactation period (if the serum pregnancy test is positive, pregnancy must be excluded and confirmed after discussion with the sponsor for enrollment).
10. For male patients whose partners are women of childbearing age, they must agree to abstain from sexual activity for at least six months from the date of signing the informed consent form until the last administration of the study drug, or use effective contraceptive methods. Male patients must also agree not to donate sperm during the same period of time.
11. The patients voluntarily joined this study, signed the informed consent form and had good compliance.

Exclusion Criteria:

1. Accompanied by untreated or active central nervous system (CNS) tumor metastasis. Subjects with a history of meningeal metastasis or those currently having meningeal metastasis.
2. Patients with other malignant tumors, excluding fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, ductal carcinoma in situ after radical resection, papillary thyroid carcinoma after radical resection, or those with other malignant tumors, must have at least a 3-year tumor-free period.
3. For those whose tumor lesions are judged by researchers to have a bleeding tendency, such as those whose imaging examinations during the screening period show that the subjects have: imaging evidence of tumor invasion or encirclement of large blood vessels;
4. Exclude subjects who have previously used VEGF/PD-1 (PD-L1) bispecific antibodies; Subjects who have previously received targeted therapy with TROP2, HER2 or Nectin-4, ADC, or any study drugs containing MMAE and whose treatment duration is less than 6 months should also be excluded. Subjects who had previously used bevacizumab were excluded.
5. Previously used immune checkpoint agonist therapy (such as CD137 agonists), anti-CD73 inhibitors, immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), and immune cell therapy (such as CAR-T) And other treatments targeting the tumor immune mechanism are not allowed to be enrolled.
6. It is known that there is an allergic reaction to CVL006, SKB264, T-DXd, Enfortumab Vedotin, pemetrexel or platinum-based or any excipient component of the study drug (including histidine, trehalose and polysorbide 20), or there is a history of severe allergic reaction to other monoclonal antibodies;
7. Have serious cardiovascular and cerebrovascular diseases, including but not limited to:

   1. Severe cardiac rhythm or conduction abnormalities within 6 months prior to the first use of the study drug, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, etc.
   2. Acute coronary syndrome, congestive heart failure (New York Heart Association (NYHA) cardiac function classification ≥ grade II), and aortic dissection occurred within 6 months prior to the first use of the study drug;
   3. There have been arteriovenous thrombotic events such as cerebrovascular accidents (transient ischemic attack, cerebral hemorrhage, stroke), deep vein thrombosis and pulmonary embolism, etc. within 6 months before the first use of the study drug;
   4. The left ventricular ejection fraction (LVEF) was less than 50% within 28 days prior to the first use of the study drug;
   5. The mean value of QTcF obtained from three electrocardiogram examinations at baseline 12 (or above) in the resting state, with QTcF> 470 ms (for females) or QTcF> 450 ms (for males);
8. There is uncontrollable pleural effusion, peritoneal effusion or pericardial effusion;
9. Patients with known or suspected interstitial pneumonia; Within three months prior to the first administration, there are other severe pulmonary diseases that seriously affect respiratory function, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia/obliterative bronchiolitis; Non-infectious pulmonary inflammation that currently requires steroid treatment;
10. Patients who have previously received immunotherapy and have developed grade ≥3 irAE or grade ≥2 immune-related myocarditis;
11. Patients with active or previous autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.) are excluded, except for those with clinically stable autoimmune thyroid diseases and type 1 diabetes.
12. Had received systemic glucocorticoids (prednisone > 10mg/ day or equivalent doses of similar drugs) or other immunosuppressants within 14 days prior to the first use of the study drug; Except for the following situations: treatment with topical, ocular, intra-articular, intranasal and inhaled glucocorticoids; Short-term use of glucocorticoids for preventive treatment (such as to prevent contrast agent allergy).
13. Within 6 months prior to the first administration, there was a history of esophageal and gastric varices, severe ulcers, unhealed wounds, abdominal fistulas, abdominal abscesses or acute gastrointestinal bleeding; A history of gastrointestinal perforation and/or fistula within 6 months prior to the first administration, severe gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), and extensive intestinal resection (partial colectomy or extensive small intestine resection);
14. Arm2.3 Exclude primary peritoneal, pericardial and testicular sheath mesothelioma.
15. Patients with Arm2.9 urothelial carcinoma, except for those with eye diseases or symptoms that may increase the risk of corneal epithelial damage before the first treatment with the study drug and are not suitable for participation in this study; Patients with a history of grade ≥2 peripheral neuropathy are excluded. Patients with baseline HbA1c≥8% were excluded.
16. There was a severe infection within 4 weeks before the start of the study treatment, including but not limited to bacteremia, severe pneumonia or other serious infectious complications that require hospitalization, etc. There is an active infection of CTCAE grade ≥ 2 that requires intravenous anti-infective treatment within 2 weeks before the first administration.
17. Have a history of immune deficiency, including a positive HIV test; There is active hepatitis B (HBV DNA higher than the upper limit of the normal value of the testing center) or hepatitis C (anti-HCV positive and HCV RNA higher than the detection limit of the analytical method);
18. Those who were found to have had active pulmonary tuberculosis infection within one year prior to enrollment through medical history or CT examination, or those with a history of active pulmonary tuberculosis infection more than one year ago but have not received regular treatment;

19. The adverse reactions of previous anti-tumor treatment have not yet recovered to CTCAE v 5.0 grade evaluation ≤1 (alopecia, grade 2 peripheral neurotoxicity (Arm2.9 requirement ≤1), except for the numerical requirements in the inclusion criteria or other situations determined by the investigator that do not affect the treatment of the study drug);

20) Those who have received chemotherapy within 3 weeks before the first use of the study drug, or have received anti-tumor treatments such as macromolecular biological therapy (including immunotherapy) or other unmarketed clinical research drugs within 4 weeks before the first use; Excluding the following items:

For oral fluorouracil and small molecule targeted drugs, it is within two weeks before the first use of the study drug or within five half-lives of the drug, whichever is shorter.

b. For traditional Chinese medicines with anti-tumor indications, it is two weeks before the first use of the study drug;

c. Radical radiotherapy is 4 weeks before the first use of the study drug, and palliative radiotherapy is 2 weeks before the first use of the study drug.

21) Having undergone major organ surgery, experienced significant trauma, or required elective surgery during the trial period within 4 weeks prior to the first use of the study drug; Perform a coarse needle biopsy or other minor surgery (excluding central venous intubation and port implantation) within 7 days before the first administration of the drug;

22. There is a history of bleeding tendency or coagulation disorder and/or clinically significant bleeding symptoms or risks within 4 weeks prior to the first administration, including but not limited to: a. Gastrointestinal bleeding b. Hemoptysis (coughing up ≥15ml of fresh blood or blood clots); c. Epistaxis/nosebleeds d. Receive therapeutic anticoagulant therapy before the first administration;

23) A history of hypertensive crisis or hypertensive encephalopathy in the past; There was hypertension within one month before the first administration and the systolic blood pressure was ≥150mmHg or the diastolic blood pressure was ≥100mmHg after oral antihypertensive drugs.

24) Active or with a previous history of inflammatory bowel disease (such as Crohn's disease, ulcerative colitis or chronic diarrhea);

25) There is a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;

26) Those who need to use strong suppressors or inducers of cytochrome P450 3A4 (CYP3A4) within 2 weeks before the first administration and during the study period (the use of strong suppressors or inducers of CYP3A4 is not allowed. The representative drugs of strong suppressors or inducers of CYP3A4 are listed in the attachment);

27) Receive a live virus vaccine 30 days before the first administration, or plan to receive a live vaccine during the study period;

28) As determined by the researchers, the subjects have other factors that may affect the research results or lead to the forced termination of this study, such as alcohol abuse, drug abuse, suffering from other serious diseases (including mental disorders) requiring concurrent treatment, severely abnormal laboratory test values, family or social factors, and other circumstances that may affect the safety of the subjects or the collection of experimental data, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2028-08-12 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
DLT and RP2D of phase I | 28 days after the first medication; If the second administration is delayed, the DLT observation period will be extended to 14 days after the second administration
  DLT and RP2D of phase I (Arm1.1, Arm1.2, Arm1.3 and Arm1.4) CVL006 combined with pemetrexed + carboplatin/SKB264/ DS-8201a/ Enfortumab Vedotin in patients with advanced solid tumors
Phase II, progression-free survival (PFS) according to RECISTv1.1 criteria | Imaging examinations should be conducted every 8 weeks (±7 days) after the initiation of administration
  The efficacy of phase II CVL006 combined with pemetrexed + carboplatin /SKB264/ DS-8201a/ Enfortumab Vedotin in the treatment of advanced solid tumors: progression-free survival (PFS) according to RECISTv1.1 criteria
Safety endpoints for phase I and Phase II | From date of randomization until the date of first documented progression, assessed up to 36 months
  Number of participants with adverse events (AE)/serious adverse events (SAE)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of CVL006 in Phase I and Phase II | From date of randomization until the date of first documented progression, assessed up to 36 months
  The pharmacokinetic (PK) parameters of CVL006 in phase I and Phase II, including but not limited to: Cmax
Pharmacokinetic (PK) parameters of CVL006 in Phase I and Phase II | From date of randomization until the date of first documented progression, assessed up to 36 months
  The pharmacokinetic (PK) parameters of CVL006 in phase I and Phase II, including but not limited to: Tmax
Efficacy endpoints for Phase I and Phase II | From date of randomization until the date of first documented progression, assessed up to 36 months
  Efficacy endpoints for Phase I and Phase II: Evaluated by the investigators based on RECISTv1.1 criteria, including objective response rate (ORR)
Efficacy endpoints for Phase I and Phase II | From date of randomization until the date of first documented progression, assessed up to 36 months
  Efficacy endpoints for Phase I and Phase II: Evaluated by the investigators based on RECISTv1.1 criteria, including Overall survival (OS)
ADA&Nab | From date of randomization until the date of first documented progression, assessed up to 36 months
  The levels of anti-drug antibody (ADA) and neutralizing antibody (Nab) of CVL006
PD-L1 expression | From date of randomization until the date of first documented progression, assessed up to 36 months
  The correlation between PD-L1 expression and response in the tumor tissues of the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No